CLINICAL TRIAL: NCT03599284
Title: The Efficacy, Safety and Pharmacokinetic of Antiplatelet Therapy for Vicagrel in Patients With Coronary Atherosclerotic Heart Disease and Planned Percutaneous Coronary Intervention: a Multi-center, Randomized, Double-blind, Triple-dummy , Parallel-controlled, Dose-exploration Phase II Trial
Brief Title: The Efficacy, Safety and Pharmacokinetic of Antiplatelet Therapy for Vicagrel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCP1-Ⅱ-01
Record Dates: First submitted 2018-07-09; First posted 2018-07-26 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Coronary Artery Disease | interventions — methyl 2-(2-acetoxy-6,7-dihydrothieno(3,2-c)pyridin-5(4H)-yl)-2-(2-chlorophenyl)acetate; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (Experimental): Experimental group 1: Vicagrel 20mg loading followed by 5mg/day for 28 days
  Interventions: Drug: Vicagrel 5mg
- Experimental group 2 (Experimental): Experimental group 2: Vicagrel 24mg loading followed by 6mg/day for 28 days
  Interventions: Drug: Vicagrel 6mg
- Experimental group 3 (Experimental): Experimental group 3: Vicagrel 30mg loading followed by 7.5mg/day for 28 days
  Interventions: Drug: Vicagrel 7.5mg
- Control group (Active Comparator): Control group: Clopidogrel 300mg loading followed by 75mg/day for 28 days
  Interventions: Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Vicagrel 5mg — Experimental group 1 : Vicagrel 20mg loading followed by 5mg/day for 28 days
  Arms: Experimental group 1
Drug: Vicagrel 6mg — Experimental group 2 : Vicagrel 24mg loading followed by 6mg/day for 28 days
  Arms: Experimental group 2
Drug: Vicagrel 7.5mg — Experimental group 3 : Vicagrel 30mg loading followed by 7.5mg/day for 28 days
  Arms: Experimental group 3
Drug: Clopidogrel 75mg — Control group : Clopidogrel 300mg loading followed by 75mg/day for 28 days
  Arms: Control group

SUMMARY:
This is a multi-center, randomized, double-blind, triple-dummy, parallel-controled, dose-exploration phase II trial. Patients with coronary atherosclerotic heart disease and planned percutaneous coronary intervention （PCI） will be randomized after informed consent, in a 1:1:1:1 ratio to the following treatment groups: Experimental group 1 : Vicagrel 20mg loading followed by 5mg/day for 28 days; Experimental group 2 : Vicagrel 24mg loading followed by 6mg/day for 28 days; Experimental group 3 : Vicagrel 30mg loading followed by 7.5mg/day for 28 days; Control group : Clopidogrel 300mg loading followed by 75mg/day for 28 days. The primary purpose of this trial is to evaluate the efficacy, safety of vicagrel antiplatelet therapy and explore dose in patients with coronary atherosclerotic heart disease during and after PCI compared with clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18-75.
* Weight ≥ 50 kg
* Patients with coronary atherosclerotic heart disease diagnosed clinically and planned percutaneous coronary intervention
* Patients with ability and willingness to sign informed consent and adherence to trial protocol.

Exclusion Criteria:

* Hemorrhagic symptoms (such as hematemesis, melena, severe or recurrent epistaxis, hemoptysis, marked hematuria, gastrointestinal bleeding, or intracranial hemorrhage), or suspected vascular malformations (such as aneurysms), or abnormal bleeding history (such as abnormal hemorrhage attributed to tooth extraction), himself or his immediate family with coagulation or bleeding disorders (such as hemophilia);
* Non-ST-segment elevation acute coronary syndrome (<2h emergency PCI), or ST-segment elevation myocardial infarction within 7 days;
* Patients with suspected aortic dissection;
* Patients with negative coronary Computed Tomography angiography（CTA）(coronary CTA depending on investigator);
* Patients with severe disease and life expectancy <1 year;
* Patients with acute peptic ulcer;
* History of hemorrhagic stroke or history of ischemic stroke within 6 months before screening and a definite diagnosis of structural abnormalities in the central nervous system;
* Patients with uncontrolled high blood pressure (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg) after drug treatment during screening;
* One of the following conditions: cardiogenic shock, chronic congestive heart with failure New York Heart Association (NYHA) grade ≥ III grade or left ventricular ejection fraction determined by echocardiography < 35%, hypotension (systolic pressure < 90 mmHg and or diastolic pressure < 60 mmHg), severe arrhythmias (including high-degree atrioventricular block, sick sinus syndrome, persistent ventricular tachycardia), severe pulmonary insufficiency, pulmonary embolism, and hepatic insufficiency (ALT or AST caused by non-cardiac diseases exceeding the upper limit of normal by more than 3 times), severe renal insufficiency (eGFR < 30 ml/min), cirrhosis;
* Patients Received P2Y12 receptor antagonist and Ⅱb/IIIa receptor inhibitor, oral anticoagulant (warfarin, rivaroxaban, dabigatran, etc.) within 14 days before screening;
* Prolonged cardiopulmonary resuscitation (more than 10 minutes) or severe trauma within 2 weeks before screening;
* Patients plan to undergo another surgery within 1 month after participating in this trial，or plan to undergo PCI procedure performed several times during the test (except for the end of the safety follow-up);
* History of severe allergies, non-allergic drug reactions or allergies to 2 or more drugs (including contrast agents), or known allergies to the similar drugs (clopidogrel, ticagrelor) as the study drug or contraindication of aspirin;
* Patients with mental disorders or alcohol dependence;
* Patients being receiving any experimental medicine or experimental medical devices;
* Prothrombin time (PT)> 1.3 times the upper limit of normal or international normalized ratio (INR)> 2.0;
* Platelet count (PLT) < 100×10^9/L or > 600×10^9/L;
* Hemoglobin < 10g/dL;
* Patients who cannot tolerate dual antiplatelet therapy for 28 days;
* Female of reproductive age with positive blood pregnancy test;
* Female with gestational intention or in lactation;
* Other unsuitable conditions considered by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-07-28 (Actual)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation | 28 days after treatment
  Inhibition of platelet aggregation will be assessed by Verifynow System

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui
  - Beijing Anzhen Hospital, Capital Medical Universily, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - First Affiliated Hospital of Zhongshan University, Guangzhou, Guangdong
  - First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Zhongda Hospital of Southeast University, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Second Hospital of Jilin University, Changchun, Jinin
  - the General Hospital of Shenyang Military Region of The Chinese People's Liberation Army（The General Hospital of Shenyang Military）, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Tianjin People's Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjing